CLINICAL TRIAL: NCT06355843
Title: Clinical Applications of Integrated PET/MR and PET/CT in the Diagnosis and Treatment of Prostate Cancer.
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The 68Ge/68Ga generator is currently at the end of its lifespan. We are trying to purchase new equipment, which will take about half a year.
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SXY
Record Dates: First submitted 2024-01-23; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer; Pet-ct
Keywords: PSMA; PET/MRI; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-FAPI PET/MRI scan (Experimental): 68Ga-PSMA PET/CT (PET/MR) before surgery or biopsy
  Interventions: Drug: 68Ga-PSMA

INTERVENTIONS:
Drug: 68Ga-PSMA — PSMA is located in prostate epithelial cells and is converted to a membrane-bound protein in prostate cancer, and PSMA expression is approximately 100 to 1000 times higher in prostate cancer tissue compared to normal prostate tissue. PSMA is expressed at high levels in 95% of prostate cancer patients and is upregulated in castration-resistant prostate cancer (CRPC) and metastatic prostate cancer. PSMA expression was also increased after androgen deprivation therapy (ADT). The use of positronuclide 68Ga-labelled PSMA small molecule inhibitors can be specifically combined with prostate cancer cells, and it is important for the diagnosis of prostate cancer and its metastatic foci through PET/CT and PET/MR visualisation.
  With the popularity of integrated PET/MR imaging, combining the higher resolution and morphological performance of MR imaging with the N-staging and M-staging of PET, the specificity of primary prostate cancer diagnosis can be greatly improved.

SUMMARY:
The goal of this study type: observational study (prospective study) is to study prostate cancer occurrence and recurrence, to specifically identify and localize tumor foci at the molecular level at an early stage, to evaluate the prognosis of patients, and to accurately stage not only intermediate- and high-risk prostate cancer patients with a primary diagnosis, but also detect recurrent foci in patients with biochemical recurrence, to restage those who have developed metastases, to assess tumor load, and to ultimately assist in determining the personalized treatment plans. The main question it aims to answer is whether 68Ga-PSMA PET/CT (PET/MR) examination is beneficial for assessing the

* Accurate staging of patients with intermediate- and high-risk prostate cancer at first diagnosis;
* Detecting recurrent lesions in patients with recurrent tumors for re-staging;
* Assessment of tumor load;
* Assessment of patient prognosis. Participants will sign an informed consent form, undergo 68Ga-PSMA PET/CT (PET/MR) before surgery or biopsy, and have regular follow-up after obtaining pathological results of surgical resection or puncture biopsy, 6 weeks after surgery or biopsy, and then every 3 months; the follow-up will include: blood PSA, whole-body bone imaging, etc.

DETAILED DESCRIPTION:
1. Title of research programme Clinical application of integrated PET/MR and PET/CT in the diagnosis and treatment of prostate cancer
2. Research background Prostate cancer is the most common malignant tumor of the urinary system. Current diagnostic tools for prostate cancer include serum prostate-specific antigen (PSA) test, transrectal prostate aspiration biopsy, etc. However, these tools are often invasive. When a patient's PSA rises again after radical prostatectomy for prostate cancer, conventional CT, MRI, and bone scintigraphy do not have a high detection rate (11%); Although multiparametric magnetic resonance imaging (mpMRI) is of undisputed importance in the T-staging of tumors, it has limited diagnostic accuracy when applied alone and is less sensitive in the diagnosis of local lymph node metastases. Currently, PET/CT has been gradually applied to different types and stages of prostate cancer. With the popularity of integrated PET/MR imaging, combining the higher resolution and morphological performance of MR imaging with the N-staging and M-staging of PET, the specificity of primary prostate cancer diagnosis can be greatly improved.

   Currently, the commonly used targeted tracers for PET examination of prostate cancer include 18F-fluorodeoxyglucose (18F-FDG), and 18F-/11C-acetate, etc., but their imaging effects are not up to the ideal level. PSMA is located in prostate epithelial cells and is converted to a membrane-bound protein in prostate cancer, and PSMA expression is approximately 100 to 1000 times higher in prostate cancer tissue compared to normal prostate tissue. PSMA is expressed at high levels in 95% of prostate cancer patients and is upregulated in castration-resistant prostate cancer (CRPC) and metastatic prostate cancer. PSMA expression was also increased after androgen deprivation therapy (ADT). The use of 68Ga-labelled PSMA small molecule inhibitors can be specifically combined with prostate cancer cells, and it is important for the diagnosis of prostate cancer and its metastatic foci through PET/CT and PET/MR visualization. 68Ga-PSMA 617 was first applied to prostate cancer patients in 2015, Afshar-Oromieh et al. conducted the first evaluation of the human biological distribution, radiation dose of this contrast agent and found that there was uptake in the kidney and salivary glands, and the detection rate of prostate cancer lesions was 73.7% (14/19). The best imaging results were obtained 2-3 h after injection, with an average radiation dose of about 0.021 mSv/mbq.
3. Research purpose This study is expected to be used for prostate cancer occurrence and recurrence, early specific identification and localization of tumor foci at the molecular level, and evaluation of patient prognosis. Not only can it accurately stage first-time intermediate- and high-risk prostate cancer patients, but it can also detect recurrent lesions in biochemically recurrent patients. Those who develop metastases are restaged to assess tumor load and ultimately assist in determining a personalized treatment plan.
4. Type of study design, method of randomization and level of blinding Type of study design: observational study (prospective study)
5. Diagnostic criteria for prostate cancer Confirmed by prostate puncture biopsy or surgical pathological histology; Endocrine therapy has shown significant efficacy.
6. Inclusion criteria for participants

   * 18 years ≤ 75 years of age;
   * Patients with clinical suspicion of prostate cancer;
   * No recent invasive tests or treatments were performed;
   * Blood count: leukocytes>4×109/L, neutrophils>2×109/L, haemoglobin>90g/L, platelets>100×109/L;
   * Cardiac function: left ventricular ejection fraction >50%;
   * Pulmonary function tests: FEV1 ≥1.2L, FEV1% ≥50% and DLCO ≥50%;
   * Liver function: total bilirubin <1.5 times upper limit of normal (ULN); AST and ALT <1.5 times ULN;
   * Renal function: serum creatinine ≤ 1.5 times ULN, or glomerular filtration rate > 60 ml/min;
   * Participants agreed to participate in this clinical trial and signed an informed consent form;
   * Good compliance and commitment to follow the study procedures and to cooperate in the implementation of the full study;
   * No birth plans for six months.
7. Exclusion Criteria for Participants

   * Those with severe psychiatric symptoms, or those who are too confused to cooperate with the examination;
   * Those with poor compliance.
8. Calculation of the number of cases required to achieve the desired aim of the study based on statistical principles This was an exploratory observational study and the sample size was not calculated based on statistical assumptions, and the sample size was initially determined to be 50 cases.
9. Criteria for discontinuing clinical studies, provisions for ending clinical studies (1)Significant errors in the clinical research protocol or serious deviations in the implementation of the protocol that make it difficult to assess the utility of the study; (2)The drug regulatory authority, government department or ethics committee asked to suspend or end the study; (3)Circumstances in which other researchers do not consider it appropriate to continue the study or find it difficult to do so.
10. Subject screening numbers, subject numbers, and case report forms are maintained Participant Screening Number: a 1-sequential number, e.g., 1-1 for the first participant; participant Number: a sequential number, e.g., 001 for the first participant; Case report form retention: information is entered into the CRF form by the project leader or other authorized investigator, and only medically qualified investigators are allowed to complete the original clinical assessment/safety data. Any changes made to the CRF form by the project leader or other authorized researchers after the original data has been entered need to be documented. Any modification of data that has been endorsed will require the name of the researcher or other authorized researcher who made the modification, the date of the modification, and the reason for the modification (if the change is minor).
11. Documentation of adverse events and methods of reporting serious adverse events, management measures, modalities, timing and regression of follow-up visits.

    11.1 Adverse events Adverse Event (AE) is an unfavorable medical event that occurs during a clinical trial. Clinical trial Any adverse event that occurs during the implementation should be faithfully recorded and analyzed for reasons. Both anticipated and unanticipated adverse events should be be recorded and reported truthfully. Adverse events should be included as outcome variables in the statistical analysis of clinical trials.

    11.2 Serious adverse event A serious Adverse Event (SAE) is a clinical trial event that results in death or serious deterioration of health, including fatal illness or injury, permanent defects in body structure or function, hospitalization or prolonged hospitalization, or the need for medical or surgical intervention to avoid permanent defects in body structure or function. Events that result in fetal distress, fetal death, or congenital anomalies or congenital defects.

    11.3 Reporting procedures 11.3.1 Reporting time frames In the event of AE or SAE in this clinical trial, the investigator shall immediately take appropriate therapeutic measures for the participant, notify the principal investigator, and report in writing to the appropriate authorities within 24 hours once SAE has been determined.

    11.3.2 Reporting Sector The office of the clinical trial organization to which it belongs, the sponsor, our Ethics Committee, as well as the drug supervision and management department of the province, autonomous region, and municipality directly under the central government where the clinical trial organization is located, and the competent department of health and wellness.

    11.3.3 Reporting methods If an SAE occurs, the investigator completes the Adverse Event Record Form and files the original Adverse Event Record Form in the investigator's file folder.

    11.3.4 Processing and recording When an SAE or suspected SAE occurs, the investigator immediately stops the trial and takes appropriate therapeutic measures, notifies the principal investigator and the sponsor; the principal investigator makes a judgment about the relevance of the SAE to the trial and records the occurrence, development, and treatment of the SAE in as much detail as possible on the Adverse Event Record Form, which is documented on the Case Report Form, signed and dated.

    11.3.5 follow-up If SAE is determined, the event must be followed until it appears to improve, stabilizes, or, in the judgment of the principal investigator, does not require follow-up.
12. Statistical analysis plan, definition, and selection of data sets for statistical analysis 12.1 General approach SPSS software was used for statistical analysis of data. If the data were normally distributed, they were expressed as mean ± standard deviation and compared using a two-sample t-test and one-way ANOVA. If the data were not normally distributed, they were expressed as M(P5, P95) and compared using the Mann-Whitneyu and Kruskal-WallisH rank sum tests. P<0.05 is considered a statistically significant difference.

    12.2 Analysis of primary and secondary study endpoints Survival analysis was performed using the Kaplan-Meier method to plot survival curves, and the log-rank test was used to compare survival differences between groups.
13. Data management and confidentiality of information 13.1 Data entry and modification Data entry and modification will be done by the Department of Nuclear Medicine, and data collection will be performed by clinical researchers under the supervision of the person in charge, who will be responsible for the accuracy, completeness, and timeliness of the reported data. All data should be clear to ensure accurate interpretation and to guarantee its traceability. Clinical data will be maintained in a database, which should be password-protected, and a logical proofreading process should be in place when the database is created.

    The Data Manager is responsible for reviewing and managing the entered data. In case of doubt about the existence of data, the data manager will send the appropriate query to the researcher, who will respond to the query sent by the data manager in a timely manner, and the data manager will be able to re-question the data if necessary.

    13.2 Confidentiality Program for Research Participant Information Participants' personal information follows the principle of confidentiality. The investigator will replace the participants' identifying information with a code name that does not contain his/her name.

    13.3 Confidentiality Program for Research Data
14. Quality control and quality assurance in clinical research 14.1 Conditions of research units and training of personnel The department in which the research project is located has the appropriate personnel, equipment and first aid facilities; All research participants (including doctors, nurses, and others) have received appropriate training in relation to the research and any information relevant to the conduct of the research has been passed on to the relevant personnel; All equipment has a technical inspection certificate from the technical supervision department indicating that it is in good working order; During the course of the trial study, the investigators should be relatively fixed, and for the change of investigators in the middle of the study, they should join the study after training, and the "Clinical Trial Participant Contact Form" should be changed again.

    14.2 Modifications to the pilot program Any modifications to the trial protocol that would affect the execution of the study, the purpose of the trial, the design of the trial, the number of patient cases and the flow of the trial, etc., must be submitted as amendments to the trial protocol, which must be agreed upon by the investigator and the Ethics Committee before they can be implemented.
15. Research-related ethics Participants are not paid and are responsible for some of the costs. The study was conducted in accordance with China's Measures for Ethical Review of Biomedical Research Involving Human Beings and international ethical guidelines such as the Declaration of Helsinki.
16. Methods of subject recruitment and process of obtaining informed consent Participant Recruitment Methods: Patients meeting the inclusion/exclusion criteria were referred by the Department of Nuclear Medicine for inclusion in the clinical study.

    Informed Consent Process: Informed consent should be completed before the participant agrees to participate in the study and should continue throughout the study. The informed consent form was agreed upon by the Ethics Committee and should be read and signed by the participants. The researcher will explain the research process answer questions from participants and inform participants of the possible risks and their rights. Participants may discuss with a family member or guardian before agreeing to participate. The investigator must inform participants that participation in the study is voluntary and that they may withdraw from the study at any time during the study. A copy of the informed consent form can be provided to the study participant to keep. The rights and welfare of subjects will be protected and it is emphasized that the quality of their medical care will not be compromised by refusal to participate in research.
17. Expected progress and completion dates of clinical studies 2022.4.28-2027.3.31 Screening of eligible participants, who underwent relevant examinations as arranged by the investigator; 2027.4.1-2027.9.30 Complete the statistical analysis of the experimental data.
18. Follow-up and medical measures at the end of the study Patients are followed up on a long-term basis and assistance is provided accordingly.

ELIGIBILITY:
Inclusion Criteria:

* 18 years ≤ 75 years of age;
* Patients with clinical suspicion of prostate cancer;
* No recent invasive tests or treatments were performed;
* Blood count: leukocytes>4×109/L, neutrophils>2×109/L, haemoglobin>90g/L, platelets>100×109/L;
* Cardiac function: left ventricular ejection fraction >50%;
* Pulmonary function tests: FEV1 ≥1.2L, FEV1% ≥50% and DLCO ≥50%;
* Liver function: total bilirubin <1.5 times upper limit of normal (ULN); AST and ALT <1.5 times ULN;
* Renal function: serum creatinine ≤ 1.5 times ULN, or glomerular filtration rate > 60 ml/min;
* Participants agreed to participate in this clinical trial and signed an informed consent form;
* Good compliance and commitment to follow the study procedures and to cooperate in the implementation of the full study;
* No birth plans for six months.

Exclusion Criteria:

* Those with severe psychiatric symptoms, or those who are too confused to cooperate with the examination;
* Those with poor compliance.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Measuring the value of 68Ga-PSMA PET/MRI in the diagnosis and staging of primary prostate cancer and comparing it with mp-MRI and PET/CT | up to 28 months
  68Ga-PSMA-11 PET/MRI and multiparametric MRI images of participants with suspected prostate cancer were collected and compared with 68Ga-PSMA-11 PET/MRI, 68Ga-PSMA-11 PET and multiparametric MRI for the diagnosis of prostate cancer, using histopathological findings as the "gold standard". Accuracy, sensitivity, specificity, positive and negative predictive values were calculated. The diagnostic efficacy of the three was analyzed by plotting the working characteristic curves of the subjects.
Exploring whether 68Ga-PSMA PET/MRI can be used as a method for diagnostic efficacy | up to 32 months
  68Ga-PSMA-11 PET/MRI images of prostate cancer patients were collected, and the histopathological findings were used as the "gold standard". The accuracy, sensitivity, specificity, positive predictive value, and negative predictive value of 68Ga-PSMA-11 PET/MRI for diagnosing T, N, and M stages of prostate cancer were calculated. The working characteristic curves of the subjects were plotted and their diagnostic efficacy was calculated by the area under the curve.

CONTACTS AND LOCATIONS:
Overall Officials: Huiqin Xu, Principal Investigator — The First Affiliated Hospital of Anhui Medical University
Locations (1):
- First affiliated hospital of anhui university, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No
The datasets generated during and/or analyzed during the current study are available from the corresponding author upon reasonable request.

REFERENCES:
- [Result] Pishgar F, Ebrahimi H, Saeedi Moghaddam S, Fitzmaurice C, Amini E. Global, Regional and National Burden of Prostate Cancer, 1990 to 2015: Results from the Global Burden of Disease Study 2015. J Urol. 2018 May;199(5):1224-1232. doi: 10.1016/j.juro.2017.10.044. Epub 2017 Nov 9. PMID 29129779
- [Result] Schoder H, Larson SM. Positron emission tomography for prostate, bladder, and renal cancer. Semin Nucl Med. 2004 Oct;34(4):274-92. doi: 10.1053/j.semnuclmed.2004.06.004. PMID 15493005
- [Result] Brawer MK, Ploch NR, Bigler SA. Prostate cancer tumor location as predicted by digital rectal examination transferred to ultrasound and ultrasound-guided prostate needle biopsy. J Cell Biochem Suppl. 1992;16H:74-7. doi: 10.1002/jcb.240501217. PMID 1289676
- [Result] Jadvar H. Prostate cancer: PET with 18F-FDG, 18F- or 11C-acetate, and 18F- or 11C-choline. J Nucl Med. 2011 Jan;52(1):81-9. doi: 10.2967/jnumed.110.077941. Epub 2010 Dec 13. PMID 21149473
- [Result] Choueiri TK, Dreicer R, Paciorek A, Carroll PR, Konety B. A model that predicts the probability of positive imaging in prostate cancer cases with biochemical failure after initial definitive local therapy. J Urol. 2008 Mar;179(3):906-10; discussion 910. doi: 10.1016/j.juro.2007.10.059. Epub 2008 Jan 22. PMID 18207194
- [Result] Heidenreich A, Bastian PJ, Bellmunt J, Bolla M, Joniau S, van der Kwast T, Mason M, Matveev V, Wiegel T, Zattoni F, Mottet N; European Association of Urology. EAU guidelines on prostate cancer. part 1: screening, diagnosis, and local treatment with curative intent-update 2013. Eur Urol. 2014 Jan;65(1):124-37. doi: 10.1016/j.eururo.2013.09.046. Epub 2013 Oct 6. PMID 24207135
- [Result] Barentsz JO, Weinreb JC, Verma S, Thoeny HC, Tempany CM, Shtern F, Padhani AR, Margolis D, Macura KJ, Haider MA, Cornud F, Choyke PL. Synopsis of the PI-RADS v2 Guidelines for Multiparametric Prostate Magnetic Resonance Imaging and Recommendations for Use. Eur Urol. 2016 Jan;69(1):41-9. doi: 10.1016/j.eururo.2015.08.038. Epub 2015 Sep 8. No abstract available. PMID 26361169
- [Result] Sivaraman A, Sanchez-Salas R. Re: can clinically significant prostate cancer be detected with multiparametric magnetic resonance imaging? A systematic review of the literature. Eur Urol. 2015 Oct;68(4):738. doi: 10.1016/j.eururo.2015.06.033. No abstract available. PMID 26334122
- [Result] Grivas N, Lardas M, Espinos EL, Lam TB, Rouviere O, Mottet N, van den Bergh RCN; Members of the EAU-EANM-ESTRO-ESUR-ISUP-SIOG Prostate Cancer Guidelines Panel. Prostate Cancer Detection Percentages of Repeat Biopsy in Patients with Positive Multiparametric Magnetic Resonance Imaging (Prostate Imaging Reporting and Data System/Likert 3-5) and Negative Initial Biopsy. A Mini Systematic Review. Eur Urol. 2022 Nov;82(5):452-457. doi: 10.1016/j.eururo.2022.07.025. Epub 2022 Aug 18. PMID 35985901
- [Result] Hovels AM, Heesakkers RA, Adang EM, Jager GJ, Strum S, Hoogeveen YL, Severens JL, Barentsz JO. The diagnostic accuracy of CT and MRI in the staging of pelvic lymph nodes in patients with prostate cancer: a meta-analysis. Clin Radiol. 2008 Apr;63(4):387-95. doi: 10.1016/j.crad.2007.05.022. Epub 2008 Feb 4. PMID 18325358
- [Result] Gorin MA, Rowe SP, Denmeade SR. Clinical Applications of Molecular Imaging in the Management of Prostate Cancer. PET Clin. 2017 Apr;12(2):185-192. doi: 10.1016/j.cpet.2016.11.001. Epub 2017 Jan 16. PMID 28267452
- [Result] Jani AB, Schreibmann E, Rossi PJ, Shelton J, Godette K, Nieh P, Master VA, Kucuk O, Goodman M, Halkar R, Cooper S, Chen Z, Schuster DM. Impact of 18F-Fluciclovine PET on Target Volume Definition for Postprostatectomy Salvage Radiotherapy: Initial Findings from a Randomized Trial. J Nucl Med. 2017 Mar;58(3):412-418. doi: 10.2967/jnumed.116.176057. Epub 2016 Sep 8. PMID 27609792
- [Result] Park SY, Zacharias C, Harrison C, Fan RE, Kunder C, Hatami N, Giesel F, Ghanouni P, Daniel B, Loening AM, Sonn GA, Iagaru A. Gallium 68 PSMA-11 PET/MR Imaging in Patients with Intermediate- or High-Risk Prostate Cancer. Radiology. 2018 Aug;288(2):495-505. doi: 10.1148/radiol.2018172232. Epub 2018 May 22. PMID 29786490
- [Result] Lutje S, Heskamp S, Cornelissen AS, Poeppel TD, van den Broek SA, Rosenbaum-Krumme S, Bockisch A, Gotthardt M, Rijpkema M, Boerman OC. PSMA Ligands for Radionuclide Imaging and Therapy of Prostate Cancer: Clinical Status. Theranostics. 2015 Oct 18;5(12):1388-401. doi: 10.7150/thno.13348. eCollection 2015. PMID 26681984
- [Result] Demirkol MO, Acar O, Ucar B, Ramazanoglu SR, Saglican Y, Esen T. Prostate-specific membrane antigen-based imaging in prostate cancer: impact on clinical decision making process. Prostate. 2015 May;75(7):748-57. doi: 10.1002/pros.22956. Epub 2015 Jan 18. PMID 25598074
- [Result] Liu T, Wu LY, Fulton MD, Johnson JM, Berkman CE. Prolonged androgen deprivation leads to downregulation of androgen receptor and prostate-specific membrane antigen in prostate cancer cells. Int J Oncol. 2012 Dec;41(6):2087-92. doi: 10.3892/ijo.2012.1649. Epub 2012 Oct 4. PMID 23041906
- [Result] Eder M, Schafer M, Bauder-Wust U, Hull WE, Wangler C, Mier W, Haberkorn U, Eisenhut M. 68Ga-complex lipophilicity and the targeting property of a urea-based PSMA inhibitor for PET imaging. Bioconjug Chem. 2012 Apr 18;23(4):688-97. doi: 10.1021/bc200279b. Epub 2012 Mar 13. PMID 22369515
- [Result] Weineisen M, Simecek J, Schottelius M, Schwaiger M, Wester HJ. Synthesis and preclinical evaluation of DOTAGA-conjugated PSMA ligands for functional imaging and endoradiotherapy of prostate cancer. EJNMMI Res. 2014 Dec;4(1):63. doi: 10.1186/s13550-014-0063-1. Epub 2014 Nov 25. PMID 26116124
- [Result] Benesova M, Schafer M, Bauder-Wust U, Afshar-Oromieh A, Kratochwil C, Mier W, Haberkorn U, Kopka K, Eder M. Preclinical Evaluation of a Tailor-Made DOTA-Conjugated PSMA Inhibitor with Optimized Linker Moiety for Imaging and Endoradiotherapy of Prostate Cancer. J Nucl Med. 2015 Jun;56(6):914-20. doi: 10.2967/jnumed.114.147413. Epub 2015 Apr 16. PMID 25883127
- [Result] Afshar-Oromieh A, Zechmann CM, Malcher A, Eder M, Eisenhut M, Linhart HG, Holland-Letz T, Hadaschik BA, Giesel FL, Debus J, Haberkorn U. Comparison of PET imaging with a (68)Ga-labelled PSMA ligand and (18)F-choline-based PET/CT for the diagnosis of recurrent prostate cancer. Eur J Nucl Med Mol Imaging. 2014 Jan;41(1):11-20. doi: 10.1007/s00259-013-2525-5. Epub 2013 Sep 27. PMID 24072344
- [Result] Afshar-Oromieh A, Hetzheim H, Kratochwil C, Benesova M, Eder M, Neels OC, Eisenhut M, Kubler W, Holland-Letz T, Giesel FL, Mier W, Kopka K, Haberkorn U. The Theranostic PSMA Ligand PSMA-617 in the Diagnosis of Prostate Cancer by PET/CT: Biodistribution in Humans, Radiation Dosimetry, and First Evaluation of Tumor Lesions. J Nucl Med. 2015 Nov;56(11):1697-705. doi: 10.2967/jnumed.115.161299. Epub 2015 Aug 20. PMID 26294298
- See also: Global, Regional and National Burden of Prostate Cancer, 1990 to 2015: Results from the Global Burden of Disease Study 2015 — https://pubmed.ncbi.nlm.nih.gov/29129779/
- See also: Positron emission tomography for prostate, bladder, and renal cancer — https://pubmed.ncbi.nlm.nih.gov/15493005/
- See also: Prostate cancer tumor location as predicted by digital rectal examination transferred to ultrasound and ultrasound-guided prostate needle biopsy — https://pubmed.ncbi.nlm.nih.gov/1289676/
- See also: Prostate cancer: PET with 18F-FDG, 18F- or 11C-acetate, and 18F- or 11C-choline — https://pubmed.ncbi.nlm.nih.gov/21149473/
- See also: A model that predicts the probability of positive imaging in prostate cancer cases with biochemical failure after initial definitive local therapy — https://pubmed.ncbi.nlm.nih.gov/18207194/
- See also: EAU guidelines on prostate cancer. part 1: screening, diagnosis, and local treatment with curative intent-update 2013 — https://pubmed.ncbi.nlm.nih.gov/24207135/
- See also: Synopsis of the PI-RADS v2 Guidelines for Multiparametric Prostate Magnetic Resonance Imaging and Recommendations for Use — https://pubmed.ncbi.nlm.nih.gov/26361169/
- See also: Re: can clinically significant prostate cancer be detected with multiparametric magnetic resonance imaging? A systematic review of the literature — https://pubmed.ncbi.nlm.nih.gov/26334122/
- See also: The diagnostic accuracy of CT and MRI in the staging of pelvic lymph nodes in patients with prostate cancer: a meta-analysis — https://pubmed.ncbi.nlm.nih.gov/18325358/
- See also: Clinical Applications of Molecular Imaging in the Management of Prostate Cancer — https://pubmed.ncbi.nlm.nih.gov/28267452/
- See also: Impact of 18F-Fluciclovine PET on Target Volume Definition for Postprostatectomy Salvage Radiotherapy: Initial Findings from a Randomized Trial — https://pubmed.ncbi.nlm.nih.gov/27609792/
- See also: Gallium 68 PSMA-11 PET/MR Imaging in Patients with Intermediate- or High-Risk Prostate Cancer — https://pubmed.ncbi.nlm.nih.gov/29786490/
- See also: PSMA Ligands for Radionuclide Imaging and Therapy of Prostate Cancer: Clinical Status — https://pubmed.ncbi.nlm.nih.gov/26681984/
- See also: Prostate-specific membrane antigen-based imaging in prostate cancer: impact on clinical decision making process — https://pubmed.ncbi.nlm.nih.gov/25598074/
- See also: Prolonged androgen deprivation leads to downregulation of androgen receptor and prostate-specific membrane antigen in prostate cancer cells — https://pubmed.ncbi.nlm.nih.gov/23041906/
- See also: 68Ga-complex lipophilicity and the targeting property of a urea-based PSMA inhibitor for PET imaging — https://pubmed.ncbi.nlm.nih.gov/22369515/
- See also: Synthesis and preclinical evaluation of DOTAGA-conjugated PSMA ligands for functional imaging and endoradiotherapy of prostate cancer — https://pubmed.ncbi.nlm.nih.gov/26116124/
- See also: Preclinical Evaluation of a Tailor-Made DOTA-Conjugated PSMA Inhibitor with Optimized Linker Moiety for Imaging and Endoradiotherapy of Prostate Cancer — https://pubmed.ncbi.nlm.nih.gov/25883127/
- See also: Comparison of PET imaging with a (68)Ga-labelled PSMA ligand and (18)F-choline-based PET/CT for the diagnosis of recurrent prostate cancer — https://pubmed.ncbi.nlm.nih.gov/24072344/
- See also: The Theranostic PSMA Ligand PSMA-617 in the Diagnosis of Prostate Cancer by PET/CT: Biodistribution in Humans, Radiation Dosimetry, and First Evaluation of Tumor Lesions — https://pubmed.ncbi.nlm.nih.gov/26294298/